CLINICAL TRIAL: NCT04306432
Title: Cognitive Function After Radiation Therapy for Primary Brain Tumours
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: DNOG-2
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-05

CONDITIONS: Primary Brain Tumour; Radiation Toxicity; Cognitive Impairment
Keywords: Brain tumour; Radiation therapy; Cognitive function; Hippocampus; Patient reported outcomes
MeSH Terms: conditions — Radiation Injuries; Cognitive Dysfunction; Brain Neoplasms | interventions — Neuropsychological Tests; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cognitive tests and Patient Reported Outcomes — Each patient will undergo cognitive tests and questionnaires

SUMMARY:
This study will assess cognitive function in patients with a primary brain tumour treated with radiation therapy (RT) to generate radio-sensitivity and volume effect parameters for the development of cognitive dysfunction. All types of brain tumours apart from glioblastoma will be included.

DETAILED DESCRIPTION:
RT is fundamental in the treatment of primary brain tumours. RT contributes to improved local control and prolonged progression-free survival in patients with a broad range of tumour types. Irradiation to the normal brain may lead to cognitive impairments. Clarifying the nature and severity of impairment in adult RT-treated brain tumour patients, including region-specific effects, are important for optimal utilization of novel conformal RT technologies such as proton therapy.

The study is a prospective nationwide study including approximately 300 brain tumour patients from the Danish Center of Particle Therapy and the four Neuro Oncology Centers in Denmark.

The patients will be assessed with a comprehensive battery of standardized cognitive tests and complete a questionnaire (PRO's). They will do this prior to RT treatment and 1, 3, 5 and 10 years afterwards. The PRO's includes measures on quality of life, fatigue, sleep, depression, anxiety, and socio demographics. The standardized tests are: Trail making Test (TMT); Hopkins Verbal Learning Test (HVLT); Controlled Oral Word Association Test (COWAT) - Animals and S; Coding and Digit Span from WAIS-IV. The correlation between cognitive scores and RT dose-volume parameters to specific areas in the brain will be tested.

This study will elucidate the dose-response relationship in radiation-induced damage to substructures of the brain such as hippocampus, thalamus, temporal and frontal lobes that will allow the clinician to prioritize these structures in planning of proton radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and Danish speaking.
* Performance status WHO 0-2
* Capable of cooperating on testing
* Tumour histology (WHO 2016 classification) of the following types: anaplastic astrocytoma (IDH mutant), diffuse astrocytoma (IDH-mutant), gemistocytic astrocytoma (IDH mutant), diffuse astrocytoma (NOS), oligodendroglioma, meningioma, medulloblastoma (NOS), pituitary adenoma, other brain tumours including skull base sarcomas

Exclusion Criteria:

* Glioblastoma
* Performance status 3-4 (Karnofsky Performances of 60 or less)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be diagnosed with a primary brain tumour and referred to radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2034-03-31 (Estimated); Study Completion 2034-03-31 (Estimated)

PRIMARY OUTCOMES:
Impairment of verbal learning and memory as assessed by the HVLT-r test | 10 Years
  Examined by the Hopkins Verbal Learning Test revised. It will be correlated to the mean radiation dose to the hippocampus. Outcome is number of correct words (0-24)

SECONDARY OUTCOMES:
Processing speed I | 10 years
  Examined by the Trail making Test part A (TMT_A). Outcome for TMT_A is time in seconds (0-120 seconds).
Processing speed II | 10 years
  Examined by the Coding from Wechsler Adult Intelligence Scale (WAIS-IV). Outcome for Coding is number of correct (within 2 minutes) (0-100)
Attention and working memory | 10 years
  Examined by Wechsler Adult Intelligence Scale (WAIS_IV_digit_span). Outcome on WAIS digit span is number of correct (0-36)
Verbal learning and memory | 10 years
  Examine by the Hopkins Verbal Learning Test revised (HVLT-r) - total and delayed. Outcome is number of correct words (0-24)
Verbal fluency | 10 years
  Examined by the Controlled Oral Word Association Test (COWAT) - Animals and letter_S. Outcome is number of words produced in 1 minute (0-100)
Executive function I | 10 years
  Examined by Trail making Test part B (TMT_B). Outcome for TMT_B is time in seconds (0-300).
Executive function II | 10 years
  Examined by the STROOP colour and word test (STROOP). Outcome for STROOP is number of corrects (0-120)
Global Health - Quality of life | 10 years
  Assessed by questionnaire; European organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) in order to examine the level of quality of life in brain tumour patients who has received radiation therapy. The total score is a number (0-100)
Side effects to radiation therapy | 10 years
  Assessed by EORTC Brain Neoplasm Questionnaire, BN20 (an addition to QLQ-C30 mentioned above) in order to measure side effects to radiation therapy for a brain tumour. the score is a number (0-100)
Quality of Sleep | 10 years
  Assessed by questionnaire: Pittsburgh Sleep Quality INDEX, (PSQI) in order to explore the level of quality of sleep in brain tumour patients who has received radiation therapy. Outcome is a number (0-33)
Fatigue | 10 years
  Assessed by questionnaire: Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue scale (version 4) in order to explore the level of fatigue in brain tumour patients who has received radiation therapy. Outcome is a number (0-52)
Depression/Anxiety | 10 years
  Assessed by questionnaire: Hospital anxiety and depression Scale (HADS) in order to explore level of depression and anxiety in patients treated with radiation therapy for their brain tumour. Outcome is a number (0-56)
Patient's Assessment of Own Functioning | 10 years
  Assessed by questionnaire; Patient's Assessment of Own Functioning Inventory (PAOFI), in order to assess patients own perception of cognitive function. Outcome is a number (35-210)

CONTACTS AND LOCATIONS:
Overall Officials: Lene Haldbo-Classen, M.D, Principal Investigator — Aarhus University Hospital
Locations (5):
- Denmark (5):
  - Department of Oncology, Rigshospitalet, Copenhagen, Capital Region
  - Danish Center for Particel Therapy, Aarhus, Region Midt
  - Department of Oncology, Aarhus University Hospital, Aarhus, Region Midt
  - Department of Oncology, Aalborg University Hospital, Aalborg, Region Nord
  - Department of Oncology, Odense University Hospital, Odense, Region Syd

IPD SHARING:
Plan to Share IPD: No